CLINICAL TRIAL: NCT00114348
Title: ALL-REZ BFM 2002: Protocol for the Treatment of Children With Relapsed Acute Lymphoblastic Leukemia
Brief Title: ALL-REZ BFM 2002: Multi-Center Study for Children With Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Kinderkrebsstiftung (Other)
Responsible Party: Principal Investigator, Gunter Henze, Clinic director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2002/6a
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoblastic Leukemia, Acute; Lymphoma, Non-Hodgkin
Keywords: non-B ALL; relapse; treatment; Relapsed non-B ALL or non-B non-Hodgkin lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Recurrence

ARMS (2):
- R-Blöcke (Active Comparator): Blocktherapie
  Interventions: Procedure: R-Blocks
- Prot-II-Ida (Experimental): a
  Interventions: Procedure: Protocol II-Ida

INTERVENTIONS:
Procedure: R-Blocks
  Arms: R-Blöcke
Procedure: Protocol II-Ida
  Arms: Prot-II-Ida

SUMMARY:
The protocol ALL-REZ BFM 2002 aims at the optimization of treatment for children with relapsed acute lymphoblastic leukemia. The primary objective of study ALL-REZ BFM 2002 is the randomized comparison of a lower dosed and less intensive, but continuous consolidation therapy with conventional therapy administered in treatment blocks. Outcome measures are the reduction of minimal residual disease (MRD), event-free and overall survival, and the toxicity associated with each treatment strategy.

DETAILED DESCRIPTION:
The study is based on the results of five consecutive trials performed by the ALL-REZ BFM study group since 1983. Thus the study meets the criteria of evidence-based therapy, which has been developed over nearly 20 years. Multi-agent chemotherapy in short intensive courses, which are separated by treatment-free intervals, has proved to be a successful form of induction and consolidation therapy. It is followed by preventative (or therapeutic) cranial irradiation and continuation therapy. A number of risk factors, particularly the time of relapse, site of relapse, and the ALL immunophenotype, allow the stratification of patients into a group that has an acceptable prognosis after treatment with chemotherapy alone and a second group that has a high risk of subsequent recurrence following the achievement of a second remission. The latter group requires further intensification of consolidation therapy by allogenic stem cell transplantation (SCT). To date, the indication for SCT has remained unclear for a large and heterogeneous group of patients with an intermediate prognosis. During the precursor study ALL-REZ BFM 96, however, the amount of minimal residual disease (MRD) determined quantitatively with clonal molecular markers after the second induction therapy element was shown to be a highly significant predictor of relapse-free survival.

The primary objective of study ALL-REZ BFM 2002 is the randomized comparison of a lower dosed and less intensive, but continuous consolidation therapy with conventional therapy administered in treatment blocks. Outcome measures are the reduction of MRD, event-free and overall survival, and the toxicity associated with each treatment strategy.

The secondary objectives include an improvement of the prognosis in the intermediate risk group using the stratification in treatment arms with and without allogenic SCT based on the MRD result after the second treatment element of induction therapy. An additional aim is to improve the remission induction rate in all groups by increasing the treatment intensity during induction. This is achieved by shortening the intervals between treatment blocks in keeping with the principles of guiding therapy as defined in the protocol. A series of biological companion studies aims to advance our understanding of the disorder and to establish novel prognostic factors that will allow a risk-adapted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Up to 18 years of age
* Morphologically confirmed diagnosis of relapsed non-B ALL or non-B non-Hodgkin lymphoma

Exclusion Criteria:

* They have completed the 18th year of life at the time the relapse is diagnosed.
* Curative therapy is declined either by patient himself/herself or the respective legal guardian
* The patient is pregnant
* The patient is breast feeding
* Essential parts of the relapse therapy are declined either by the patient or his/her legal cannot be administered because of medical reasons.
* No consent is given for transmission of data
* The patient has a severe concomitant disease that does not allow treatment according to protocol (e.g. malformation syndromes, cardiac malformations, metabolic disorders).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 338 (Actual)
Dates: Start 2003-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reduction of MRD | a
event-free and overall survival | a
the toxicity associated with each treatment strategy | a

SECONDARY OUTCOMES:
Improvement of the prognosis in the intermediate risk group using the stratification in treatment arms with and without allogenic SCT based on the MRD result after the second treatment element of induction therapy | a

CONTACTS AND LOCATIONS:
Overall Officials: Günter Henze, Prof.Dr.med., Principal Investigator — German Society for Pediatric Oncology and Hematology GPOH gGmbH
Locations (1):
- ALL-REZ Studienzentrale, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Taube T, Eckert C, Korner G, Henze G, Seeger K. Real-time quantification of TEL-AML1 fusion transcripts for MRD detection in relapsed childhood acute lymphoblastic leukaemia. Comparison with antigen receptor-based MRD quantification methods. Leuk Res. 2004 Jul;28(7):699-706. doi: 10.1016/j.leukres.2003.11.006. PMID 15158091
- [Result] Eckert C, Einsiedel HG, Hartmann R, von Stackelberg A, Volpel S, Guggemos A, Hanzsch N, Kawan L, Seeger K, Henze G. Clonal stability of initial leukemia in a child with central nervous system relapse 7.4 years after bone marrow relapse of common acute lymphoblastic leukemic. Haematologica. 2004 Jul;89(7):ECR23. PMID 15257960
- [Result] Wellmann S, Guschmann M, Griethe W, Eckert C, von Stackelberg A, Lottaz C, Moderegger E, Einsiedel HG, Eckardt KU, Henze G, Seeger K. Activation of the HIF pathway in childhood ALL, prognostic implications of VEGF. Leukemia. 2004 May;18(5):926-33. doi: 10.1038/sj.leu.2403332. PMID 15014526
- [Result] Herold R, von Stackelberg A, Hartmann R, Eisenreich B, Henze G. Acute lymphoblastic leukemia-relapse study of the Berlin-Frankfurt-Munster Group (ALL-REZ BFM) experience: early treatment intensity makes the difference. J Clin Oncol. 2004 Feb 1;22(3):569-70; author reply 570-1. doi: 10.1200/JCO.2004.99.153. No abstract available. PMID 14752084
- [Derived] Eckert C, Parker C, Moorman AV, Irving JA, Kirschner-Schwabe R, Groeneveld-Krentz S, Revesz T, Hoogerbrugge P, Hancock J, Sutton R, Henze G, Chen-Santel C, Attarbaschi A, Bourquin JP, Sramkova L, Zimmermann M, Krishnan S, von Stackelberg A, Saha V. Risk factors and outcomes in children with high-risk B-cell precursor and T-cell relapsed acute lymphoblastic leukaemia: combined analysis of ALLR3 and ALL-REZ BFM 2002 clinical trials. Eur J Cancer. 2021 Jul;151:175-189. doi: 10.1016/j.ejca.2021.03.034. Epub 2021 May 16. PMID 34010787
- [Derived] Eckert C, Groeneveld-Krentz S, Kirschner-Schwabe R, Hagedorn N, Chen-Santel C, Bader P, Borkhardt A, Cario G, Escherich G, Panzer-Grumayer R, Astrahantseff K, Eggert A, Sramkova L, Attarbaschi A, Bourquin JP, Peters C, Henze G, von Stackelberg A; ALL-REZ BFM Trial Group. Improving Stratification for Children With Late Bone Marrow B-Cell Acute Lymphoblastic Leukemia Relapses With Refined Response Classification and Integration of Genetics. J Clin Oncol. 2019 Dec 20;37(36):3493-3506. doi: 10.1200/JCO.19.01694. Epub 2019 Oct 23. PMID 31644328
- [Derived] Karawajew L, Dworzak M, Ratei R, Rhein P, Gaipa G, Buldini B, Basso G, Hrusak O, Ludwig WD, Henze G, Seeger K, von Stackelberg A, Mejstrikova E, Eckert C. Minimal residual disease analysis by eight-color flow cytometry in relapsed childhood acute lymphoblastic leukemia. Haematologica. 2015 Jul;100(7):935-44. doi: 10.3324/haematol.2014.116707. Epub 2015 May 22. PMID 26001791
- [Derived] Irving J, Matheson E, Minto L, Blair H, Case M, Halsey C, Swidenbank I, Ponthan F, Kirschner-Schwabe R, Groeneveld-Krentz S, Hof J, Allan J, Harrison C, Vormoor J, von Stackelberg A, Eckert C. Ras pathway mutations are prevalent in relapsed childhood acute lymphoblastic leukemia and confer sensitivity to MEK inhibition. Blood. 2014 Nov 27;124(23):3420-30. doi: 10.1182/blood-2014-04-531871. Epub 2014 Sep 24. PMID 25253770
- [Derived] Eckert C, Henze G, Seeger K, Hagedorn N, Mann G, Panzer-Grumayer R, Peters C, Klingebiel T, Borkhardt A, Schrappe M, Schrauder A, Escherich G, Sramkova L, Niggli F, Hitzler J, von Stackelberg A. Use of allogeneic hematopoietic stem-cell transplantation based on minimal residual disease response improves outcomes for children with relapsed acute lymphoblastic leukemia in the intermediate-risk group. J Clin Oncol. 2013 Jul 20;31(21):2736-42. doi: 10.1200/JCO.2012.48.5680. Epub 2013 Jun 17. PMID 23775972
- [Derived] Willer A, Gerss J, Konig T, Franke D, Kuhnel HJ, Henze G, von Stackelberg A, Moricke A, Schrappe M, Boos J, Lanvers-Kaminsky C. Anti-Escherichia coli asparaginase antibody levels determine the activity of second-line treatment with pegylated E coli asparaginase: a retrospective analysis within the ALL-BFM trials. Blood. 2011 Nov 24;118(22):5774-82. doi: 10.1182/blood-2011-07-367904. Epub 2011 Sep 22. PMID 21940824
- [Derived] Shalapour S, Hof J, Kirschner-Schwabe R, Bastian L, Eckert C, Prada J, Henze G, von Stackelberg A, Seeger K. High VLA-4 expression is associated with adverse outcome and distinct gene expression changes in childhood B-cell precursor acute lymphoblastic leukemia at first relapse. Haematologica. 2011 Nov;96(11):1627-35. doi: 10.3324/haematol.2011.047993. Epub 2011 Aug 9. PMID 21828124
- See also: ALL-REZ BFM 2002 — http://www.kinderkrebsinfo.de/